CLINICAL TRIAL: NCT05658666
Title: Leren Zien Wat Werkt: Video Interventie Ouderenzorg (VIO) Bij cliënten Met Dementie en Ernstig Probleemgedrag in Verpleeghuizen.
Brief Title: Video Feedback Intervention in Nursing Home Residents With Dementia and Severe Challenging Behavior.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 111972
Record Dates: First submitted 2022-11-29; First posted 2022-12-21 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-08

CONDITIONS: Dementia; Nursing Home Resident; Challenging Behavior
Keywords: Video Feedback Intervention; Dementia; Challenging behavior; Nursing home
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Video feedback intervention (in Dutch: Video Interventie Ouderenzorg) — The video feedback trainer assesses the interaction between the person with dementia and the caregiver and acquires agreement from the caregiver on the goals of the intervention. Caregivers are trained during several feedback sessions using personal video footage of interaction between the person with dementia and the caregiver. The feedback focuses on basic interaction and attunement principles, and the team feeling competent. Recording starts with a nondemanding situation, enabling the caregiver to become aware of the principles they already apply and to learn how these principles can be used in more demanding situations. Subsequently, video footage is recorded in 1 to 3 situations, depending on the progress, of increasing difficulty, with about 4 weeks between 2 recordings. After each recording, a 1-hour feedback session is held. The intervention concludes with separate, 30-minute sessions for the formal and informal caregivers evaluating the intervention.

SUMMARY:
The purpose of this study is to evaluate how, under what circumstances and for whom the video feedback intervention works for (the caregivers of) people with dementia and severe challenging behavior in a nursing home setting.

DETAILED DESCRIPTION:
This mixed multiple case study focuses on the evaluation of a video feedback intervention for (the caregivers of) people with dementia and challenging behavior. The video feedback intervention focuses on understanding the person with dementia, increasing the sense of competence in caregivers and improving their communication skills when interacting with the person with dementia. This realist evaluation aims to investigate what outcomes the intervention generates, for whom and in which contexts. Participants will receive care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home resident
* Dementia
* Severe challenging behavior
* Video feedback intervention is started by health care professionals as part of usual care

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Nursing home residents with dementia and severe challenging behavior where video feedback intervention is started by health care professionals as part of usual care.
  * Family caregivers of these nursing home resident
  * Involded professional caregivers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in sense of competence of the professional caregiver | 5 months
  Sense of competence in dementia care scale (SCIDS)

SECONDARY OUTCOMES:
Professional caregiver measures: changes in strain in dementia work | 5 months
  Strain in dementia care scale (SDC)
Professional caregiver measures: changes in safety in team participation | 5 months
  Team climate inventory (TCI)
Loved ones measures: changes in sense of competence | 5 months
  Short sense of competence questionnaire (SSCQ)
Person with dementia: changes in frequency of psychopathology | 5 months
  Neuropsychiatric inventory nursing home (NPI-NH)
Person with dementia: changes in severity of psychopathology | 5 months
  Neuropsychiatric inventory nursing home (NPI-NH)
Person with dementia: changes in frequency of agitated behaviors | 5 months
  Cohen Mansfield Agitation Inventory (CMAI)
Person with dementia: changes in quality of life | 5 months
  Quality of life - Alzheimer Disease Scale (QOL-AD)
Person with dementia: changes in social well-being | 5 months
  Revised index for social engagement (RISE)

OTHER OUTCOMES:
Professional caregiver measures: Changes in quality of communication with the person with dementia | 5 months
  self-developed items
Professional caregiver measures: changes in quality of relationship with the person with dementia | 5 months
  self-developed items
Professional caregiver measures: changes in emotional strain | 5 months
  self-developed items
Loved ones measures: Changes in quality of communication with the person with dementia | 5 months
  self-developed items
Loved ones measures: Changes in quality of relationship with the person with dementia | 5 months
  self-developed items
Loved ones measures: Changes in emotional strain | 5 months
  self-developed items
Loved ones measures: Changes in life satisfaction | 5 months
  self-developed items
Care team measures: changes in succesful communication with the person with dementia | 5 months
  succesful communication scheme
Care team measures: changes in attunement with the person with dementia | 5 months
  relational attunement scheme
Care team measures: Changes in sense of competence of the care team as a whole | 5 months
  Analysis team learning scale

CONTACTS AND LOCATIONS:
Overall Officials: Debby Gerritsen, Principal Investigator — Radboud University Medical Center
Locations (1):
- Expertise Centrum VIO de Wever, behandelcentrum de Hazelaar, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided